CLINICAL TRIAL: NCT07341230
Title: Deep Brain Stimulation for Disorders of Addiction: Mechanisms and a Pilot Blinded Randomized Cross-over Placebo Controlled Trial
Brief Title: Deep Brain Stimulation to Understand and Treat Addiction
Acronym: Brain-PACER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Valerie Voon, Professor Valerie Voon, Professor of Neuropsychiatry and Neuromodulation, Department of Psychiatry, University of Cambridge, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A096527; MR/W020408/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2025-12-09; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol use disorder (AUD); Deep brain stimulation (DBS); Addiction
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: This study uses a multiphase design consisting of an initial open-label optimization phase followed by a randomized, double-blind, 4-arm crossover trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dual Stimulation (Nucleus Accumbens + Ventral Internal Capsule) (Experimental): Participants receive active deep brain stimulation simultaneously targeting both the nucleus accumbens and the ventral internal capsule.
  Interventions: Device: Dual-Target Deep Brain Stimulation
- Single Stimulation - Nucleus Accumbens Only (Active Comparator): Participants receive active deep brain stimulation targeting the nucleus accumbens only, with ventral internal capsule stimulation inactive.
  Interventions: Device: Nucleus Accumbens Deep Brain Stimulation
- Single Stimulation - Ventral Internal Capsule Only (Active Comparator): Participants receive active deep brain stimulation targeting the ventral internal capsule only, with nucleus accumbens stimulation inactive.
  Interventions: Device: Ventral Internal Capsule Deep Brain Stimulation
- Sham Stimulation (Inactive) (Sham Comparator): Participants receive sham (inactive) deep brain stimulation. The implanted device is turned off; no therapeutic stimulation is provided.
  Interventions: Device: Sham Deep Brain Stimulation

INTERVENTIONS:
Device: Dual-Target Deep Brain Stimulation — A surgically implanted deep brain stimulation (DBS) system delivers active stimulation simultaneously to the nucleus accumbens and the ventral internal capsule. Stimulation parameters are based on individualized optimization performed prior to randomization and remain constant throughout this condition.
  Arms: Dual Stimulation (Nucleus Accumbens + Ventral Internal Capsule)
Device: Nucleus Accumbens Deep Brain Stimulation — A surgically implanted deep brain stimulation (DBS) system delivers active stimulation to the nucleus accumbens only. Ventral internal capsule stimulation is inactive. Stimulation parameters are based on individualized optimization performed prior to randomization and remain constant throughout this condition.
  Arms: Single Stimulation - Nucleus Accumbens Only
Device: Ventral Internal Capsule Deep Brain Stimulation — A surgically implanted deep brain stimulation (DBS) system delivers active stimulation to the ventral internal capsule only. Nucleus accumbens stimulation is inactive. Stimulation parameters are based on individualized optimization performed prior to randomization and remain constant throughout this condition.
  Arms: Single Stimulation - Ventral Internal Capsule Only
Device: Sham Deep Brain Stimulation — A surgically implanted deep brain stimulation (DBS) system is present but no therapeutic stimulation is delivered during this condition. All stimulation remains inactive.
  Arms: Sham Stimulation (Inactive)

SUMMARY:
This study is testing whether deep brain stimulation (DBS) can safely help people with severe alcohol use disorder who have not improved with standard treatments. DBS uses small electrical signals to change activity in brain areas linked to craving, self-control, and emotion. The study will test whether this treatment can reduce how often people drink and how much they drink each day. Researchers will also record brain activity to better understand how DBS affects craving and relapse.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is a leading cause of preventable illness and death worldwide and remains a major public health concern. In the United Kingdom, alcohol misuse is the greatest risk factor for death and disability among adults aged 15-49, yet many people relapse despite standard treatments. Treatment-refractory AUD therefore represents an urgent unmet clinical need. Addiction is increasingly viewed as a disorder of maladaptive brain network activity involving dysregulation of motivation, reward, stress, and executive-control systems.

Deep brain stimulation (DBS) delivers small electrical pulses to targeted brain areas to restore balanced network activity. DBS is established for movement and obsessive-compulsive disorders, and early studies suggest potential benefit for substance addictions.

This pilot trial tests dual-target DBS of the nucleus accumbens and ventral internal capsule to modulate circuits supporting craving, emotion, and self-control. Participants with severe, treatment-resistant AUD will undergo an initial open-label optimization phase followed by a randomized, blinded cross-over comparison of dual, single-site, and sham stimulation. Primary outcomes are changes in drinking frequency and quantity. Intracranial recordings from the implanted device will capture local field potentials to identify brain-signal patterns linked to craving and emotion, helping guide the development of future adaptive neuromodulation approaches for addiction.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years
* Diagnosed with Alcohol Use Disorder (AUD) according to DSM-5 criteria
* Primary diagnosis of treatment-refractory AUD (comorbid nicotine dependence, other psychoactive substance use disorders, moderate major depressive disorder, anxiety disorders or obsessive-compulsive disorder are permissible if AUD is principal)
* Disorder duration of AUD ≥ 5 years
* At least 3 unsuccessful attempts at achieving abstinence
* Failed prior psychotherapy and standard pharmacotherapy for AUD
* Medically and neurologically suitable for surgery and MRI-compatible
* Capable of providing informed consent and willing to comply with study procedures

Exclusion Criteria:

* Severe psychiatric disorder other than Alcohol Use Disorder (e.g., schizophrenia, schizoaffective disorder, bipolar disorder)
* Severe major depressive disorder (moderate depression acceptable)
* Current active suicidal ideation or history of serious suicide attempts
* Previous treatment with electroconvulsive therapy (ECT)
* Presence of implanted electrical devices, including:
* Cardiac pacemaker or defibrillator (or clinical indication for pacemaker placement)
* Implanted vagus nerve stimulator (VNS)
* Any other chronically implanted neurostimulation device
* Significant neurological history, including prior hemorrhagic or ischemic stroke, subarachnoid hemorrhage, or other major neurological illness
* Any significant medical condition that, in the opinion of the clinical team, would increase surgical or anesthetic risk
* Current pregnancy
* Contraindications to deep brain stimulation or neurosurgery, including:
* Inability to tolerate general anesthesia (as assessed by anesthesiology)
* Increased risk of bleeding (as determined by hepatology/hematology review)
* History of coagulopathy
* Current or previous anticoagulant use
* Uncontrolled hypertension (controlled hypertension with medication is acceptable)
* Stage 4 liver cirrhosis
* History of major cardiac arrhythmia (e.g., atrial fibrillation) or need for anti-arrhythmic medication
* History of requiring cardioversion
* History of repeated falls
* History of major head injury
* Marked cognitive impairment
* Seizure history, including multiple alcohol withdrawal seizures
* Marked cortical atrophy on neuroimaging

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Drinking Days per Week (Timeline Followback) | Baseline (6 months pre-surgery), monthly during open-label (Months 1-6) and randomized cross-over (Months 6-10) phases
  Alcohol use will be assessed using the Timeline Followback (TLFB), a validated self-report measure of daily alcohol consumption. Participants will report the number of days per week on which alcohol was consumed. TLFB data are collected for a 6-month pre-surgical baseline, monthly during the 6-month open-label optimization phase, and monthly during the 4-month randomized cross-over phase. Changes in drinking frequency across phases and stimulation conditions will be compared to evaluate the effect of deep brain stimulation on alcohol use.
Change in Number of Alcohol Units Consumed per Week (Timeline Followback) | Baseline (6 months pre-surgery), monthly during open-label (Months 1-6) and randomized cross-over (Months 6-10) phases
  Weekly alcohol intake will be quantified using the Timeline Followback (TLFB). The total number of standard UK alcohol units consumed per week will be calculated from participant self-report. TLFB data are collected for a 6-month pre-surgical baseline, monthly during the 6-month open-label optimization phase, and monthly during the 4-month randomized cross-over phase. Changes in total weekly consumption across phases and stimulation conditions will be compared to determine the effect of deep brain stimulation on overall drinking volume.
Adverse Events Related to Surgery or Stimulation | Continuously monitored from surgery (Day 1) through the end of Month 10 (study completion)
  All adverse events related to DBS surgery, the implanted device, or stimulation are recorded and reviewed by the clinical and research teams. Events are categorized by severity (mild, moderate, severe) and relatedness (unrelated, possibly related, related). Higher severity classifications indicate more serious adverse outcomes.

SECONDARY OUTCOMES:
Change in Alcohol Craving (Alcohol Urge Questionnaire) | Baseline (pre-surgery), daily during open-label (Months 1-6) and randomized cross-over (Months 6-10) phases
  Alcohol craving will be assessed using the Alcohol Urge Questionnaire (AUQ), a validated self-report measure of desire to drink, anticipated effects, and perceived control over drinking. Scores range from 8 to 56, with higher scores indicating stronger craving. Participants complete the AUQ daily during the open-label and randomized phases and monthly during laboratory sessions.
Quality of Life (Short Form Health Survey) | Baseline (pre-surgery), monthly during open-label (Months 1-6) and randomized cross-over (Months 6-10) phases
  Health-related quality of life will be assessed with the Short Form Health Survey (SF-36), a 36-item self-report measure comprising eight domains of physical and mental health. Domain scores are transformed to a 0-100 scale, with higher scores indicating better health status. Physical and Mental Component Summary scores may also be calculated, with higher scores reflecting better quality of life.
Illness Severity (Clinical Global Impression) | Baseline (pre-surgery), monthly during open-label (Months 1-6) and randomized cross-over (Months 6-10) phases
  Illness severity and clinical change over time will be assessed with The Clinical Global Impression (CGI) scale. The CGI-Severity (CGI-S) is a clinician-rated measure of current illness severity ranked on a 7-point scale, whereby the CGI-Improvement (CGI-I) rates change from baseline on a 7-point scale. Lower scores indicate lower severity and greater improvement.
Momentary Mood, Craving, Anxiety (0-100 VAS via WebApp) | Up to five times daily from Baseline (pre-surgery), during open-label (Months 1-6) and randomized cross-over (Months 6-10) phases
  Participants complete high-frequency ecological momentary assessments (EMAs) via a smartphone-based web application up to five times per day. Each EMA consists of composite of single-item visual analogue scale (VAS) questions assessing current depression, anxiety, and craving (e.g., "What is your craving right now?"). Responses are recorded on a continuous scale from 0 to 100, where 0 indicates none/not at all and 100 indicates the most extreme level. Higher scores indicate greater levels of the assessed state.
Cue-Induced Alcohol Craving (0-100 VAS Following Presentation of Personalized Alcohol Cues) | During perioperative laboratory testing (Days 1-7) and monthly laboratory sessions during open-label (Months 1-6) and RCT (Months 6-10) phases
  Cue-induced craving is assessed using a 0-100 visual analogue scale immediately after viewing personalized alcohol-related cues in laboratory sessions. Participants rate their urge to drink after each cue, with 0 representing "no urge" and 100 representing the "strongest imaginable urge." Higher scores indicate stronger cue-induced craving.
Daily Ecological Momentary Assessment of Depressive Symptoms (PHQ-9 Items) | Once daily from Baseline (pre-surgery), during the 6-month open-label optimization (Months 1-6) and 4-month RCT (Months 6-10) phases
  Depressive symptoms are assessed once daily using a battery comprising the nine items of the Patient Health Questionnaire-9 (PHQ-9), adapted for daily assessment. Items are administered via a smartphone-accessible Qualtrics survey and assess current depressive symptom severity. Each item is rated using a continuous visual analogue scale (VAS) ranging from 0 (not at all) to 100 (most extreme). Higher scores indicate greater depressive symptom severity.
Daily Ecological Momentary Assessment of Anxiety Symptoms (GAD-7 Items) | Once daily from Baseline (pre-surgery), during the 6-month open-label optimization (Months 1-6) and 4-month RCT (Months 6-10) phases
  Anxiety symptoms are assessed once daily using a battery comprising the seven items of the Generalized Anxiety Disorder-7 (GAD-7), adapted for daily assessment. Items are administered via a smartphone-accessible Qualtrics survey and assess current anxiety symptom severity. Each item is rated using a continuous visual analogue scale (VAS) ranging from 0 (not at all) to 100 (most extreme). Items are not rated using Likert-type response options. Higher scores indicate greater anxiety symptom severity.
Daily Ecological Momentary Assessment of Alcohol Urge (AUQ Items) | Once daily from Baseline (pre-surgery), during the 6-month open-label optimization (Months 1-6) and 4-month RCT (Months 6-10) phases
  Alcohol urge is assessed once daily using an ecological momentary assessment (EMA) battery comprising the eight items of the Alcohol Urge Questionnaire (AUQ), adapted for daily assessment. Items are administered via a smartphone-accessible survey and assess current alcohol urge. Each item is rated using a continuous visual analogue scale (VAS) ranging from 0 (no urge) to 100 (strongest urge). Items are not rated using Likert-type response options. Higher scores indicate greater alcohol urge.
Daily Assessment of Delay Discounting (Monetary Choice Questionnaire) | Once daily from Baseline (pre-surgery), during the 6-month open-label optimization (Months 1-6) and 4-month RCT (Months 6-10) phases
  Delay discounting is assessed once daily using the Monetary Choice Questionnaire (MCQ), administered via a smartphone-accessible Qualtrics survey. The MCQ comprises a series of 27 choice items in which participants select between a smaller, sooner monetary reward and a larger, later monetary reward. Each item requires a forced choice between the shorter-delay and longer-delay option. Responses are used to characterize individual differences in delay discounting, with a stronger preference for sooner rewards reflecting steeper discounting.
Daily Assessment of Risk-Taking Behavior (Mixed Gamble Task) | Once daily from Baseline (pre-surgery), during the 6-month open-label optimization (Months 1-6) and 4-month RCT (Months 6-10) phases
  Risk-taking behavior is assessed once daily using a mixed gamble decision-making task administered via an online application. On each of the 80 total trials, participants are presented with gambles offering a 50% probability of monetary gain and a 50% probability of monetary loss, with the magnitudes of potential gains and losses varying across trials. Participants indicate whether they would accept or reject each gamble. Patterns of acceptance and rejection across varying gain-loss combinations are used to characterize individual differences in risk-taking behavior, with greater acceptance of gambles indicating increased risk-taking.
Compulsive Alcohol-Related Thoughts and Behaviours (Obsessive-Compulsive Drinking Scale) | Baseline (pre-surgery) and monthly during open-label (Months 1-6) and randomized cross-over (Months 6-10) phases
  Compulsive alcohol-related thoughts and behaviors are assessed using the Obsessive-Compulsive Drinking Scale (OCDUS). Scores range from 0 to 56, with higher scores indicating more severe obsessive thoughts, urges, and loss of control related to drinking. Participants complete the OCDUS monthly to evaluate changes across study phases.
Local Field Potential (LFP) Activity During Rest and Task Performance | During perioperative phase (Days 1-7), and monthly during open-label (Months 1-6) and RCT (Months 6-10) phases
  Local field potentials (LFPs) are recorded from implanted deep brain stimulation electrodes during resting-state periods and during computerized behavioral tasks. LFP recordings are used to characterize neural activity associated with behavioral state and task performance.
Scalp Electroencephalography (EEG) Activity During Rest and Task Performance | During perioperative phase (Days 1-7), and monthly during open-label (Months 1-6) and RCT (Months 6-10) phases
  Scalp electroencephalography (EEG) is recorded during resting-state periods and during computerized behavioral tasks. EEG recordings are used to characterize cortical neural activity associated with behavioral state and task performance.
Peripheral Physiological Activity During Laboratory Task Performance | During perioperative phase (Days 1-7), and monthly during open-label (Months 1-6) and RCT (Months 6-10) phases
  Peripheral physiological signals are recorded during laboratory sessions while participants complete resting-state assessments and computerized behavioral tasks. Measures include heart rate, heart rate variability, and galvanized skin response, and are used to characterize autonomic and physiological responses associated with task performance.
Continuous Peripheral Physiological Activity During Daily Life (Wearable Monitoring) | Continuously monitored from Baseline (pre-surgery) through the end of Month 10 (study completion)
  Peripheral physiological signals are continuously recorded during daily life using a wearable device. Measures include heart rate, heart rate variability, and galvanized skin response, and are used to characterize autonomic and physiological activity over time outside the laboratory setting.
Cognitive Performance (Executive Function, Impulsivity, and Compulsivity Tasks) | Baseline (pre-surgery) and monthly during open-label (Months 1-6) and randomized cross-over (Months 6-10) phases.
  Cognitive domains including executive function, impulsivity, and compulsivity are assessed during laboratory sessions using a battery of validated computerized behavioral tasks. Tasks are designed to probe components of cognitive control, decision-making, and behavioral flexibility. Performance measures derived from these tasks are used to characterize individual differences in these cognitive domains.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals (Addenbrooke's Hospital), Cambridge, Cambridgeshire
  - King's College Hospital, London, Greater London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie published results may be shared with researchers upon reasonable request, following approval by the study investigators and institutional ethics committees. Data will be shared in accordance with relevant data protection regulations and participant consent. No personally identifiable information will be released.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 12 months after publication of primary results and for up to 5 years thereafter.
Access Criteria: Requests should be directed to the Chief Investigator (Professor Valerie Voon) via the University of Cambridge and will require a data-sharing agreement approved by the Sponsor.
URL: https://www.data.cam.ac.uk/about

REFERENCES:
- [Result] Rezai AR, Mahoney JJ, Ranjan M, Haut MW, Zheng W, Lander LR, Berry JH, Farmer DL, Marton JL, Tirumalai P, Mears A, Thompson-Lake DGY, Finomore VS, D'Haese PF, Aklin WM, George DT, Corrigan JD, Hodder SL. Safety and feasibility clinical trial of nucleus accumbens deep brain stimulation for treatment-refractory opioid use disorder. J Neurosurg. 2023 Jun 9;140(1):231-239. doi: 10.3171/2023.4.JNS23114. Print 2024 Jan 1. PMID 37329519
- [Result] Davidson B, Giacobbe P, George TP, Nestor SM, Rabin JS, Goubran M, Nyman AJ, Baskaran A, Meng Y, Pople CB, Graham SJ, Tam F, Hamani C, Lipsman N. Deep brain stimulation of the nucleus accumbens in the treatment of severe alcohol use disorder: a phase I pilot trial. Mol Psychiatry. 2022 Oct;27(10):3992-4000. doi: 10.1038/s41380-022-01677-6. Epub 2022 Jul 21. PMID 35858989
- [Result] Bach P, Luderer M, Muller UJ, Jakobs M, Baldermann JC, Voges J, Kiening K, Lux A, Visser-Vandewalle V; DeBraSTRA study group; Bogerts B, Kuhn J, Mann K. Deep brain stimulation of the nucleus accumbens in treatment-resistant alcohol use disorder: a double-blind randomized controlled multi-center trial. Transl Psychiatry. 2023 Feb 8;13(1):49. doi: 10.1038/s41398-023-02337-1. PMID 36755017
- [Result] Chen L, Li N, Ge S, Lozano AM, Lee DJ, Yang C, Li L, Bai Q, Lu H, Wang J, Wang X, Li J, Jing J, Su M, Wei L, Wang X, Gao G. Long-term results after deep brain stimulation of nucleus accumbens and the anterior limb of the internal capsule for preventing heroin relapse: An open-label pilot study. Brain Stimul. 2019 Jan-Feb;12(1):175-183. doi: 10.1016/j.brs.2018.09.006. Epub 2018 Sep 14. PMID 30245163
- [Result] Muller UJ, Voges J, Steiner J, Galazky I, Heinze HJ, Moller M, Pisapia J, Halpern C, Caplan A, Bogerts B, Kuhn J. Deep brain stimulation of the nucleus accumbens for the treatment of addiction. Ann N Y Acad Sci. 2013 Apr;1282:119-28. doi: 10.1111/j.1749-6632.2012.06834.x. Epub 2012 Dec 10. PMID 23227826
- [Result] Denys D, Mantione M, Figee M, van den Munckhof P, Koerselman F, Westenberg H, Bosch A, Schuurman R. Deep brain stimulation of the nucleus accumbens for treatment-refractory obsessive-compulsive disorder. Arch Gen Psychiatry. 2010 Oct;67(10):1061-8. doi: 10.1001/archgenpsychiatry.2010.122. PMID 20921122
- [Result] Deuschl G, Schade-Brittinger C, Krack P, Volkmann J, Schafer H, Botzel K, Daniels C, Deutschlander A, Dillmann U, Eisner W, Gruber D, Hamel W, Herzog J, Hilker R, Klebe S, Kloss M, Koy J, Krause M, Kupsch A, Lorenz D, Lorenzl S, Mehdorn HM, Moringlane JR, Oertel W, Pinsker MO, Reichmann H, Reuss A, Schneider GH, Schnitzler A, Steude U, Sturm V, Timmermann L, Tronnier V, Trottenberg T, Wojtecki L, Wolf E, Poewe W, Voges J; German Parkinson Study Group, Neurostimulation Section. A randomized trial of deep-brain stimulation for Parkinson's disease. N Engl J Med. 2006 Aug 31;355(9):896-908. doi: 10.1056/NEJMoa060281. PMID 16943402
- [Result] Voon V, Grodin E, Mandali A, Morris L, Donamayor N, Weidacker K, Kwako L, Goldman D, Koob GF, Momenan R. Addictions NeuroImaging Assessment (ANIA): Towards an integrative framework for alcohol use disorder. Neurosci Biobehav Rev. 2020 Jun;113:492-506. doi: 10.1016/j.neubiorev.2020.04.004. Epub 2020 Apr 13. PMID 32298710
- See also: Official study website for the Brain-PACER (Deep Brain Stimulation for Addictions) project, providing information about the trial, research aims, participating sites, and study team. — https://brain-pacer.com/